CLINICAL TRIAL: NCT03284008
Title: Assessing Efficacy of Axillary Web Syndrome Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Collaborators: Fondazione Umberto Veronesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IEO S721/412
Record Dates: First submitted 2017-07-25; First posted 2017-09-15 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Axillary Web Syndrome
Keywords: Breast Neoplasm; Physiotherapy; Rehabilitation
MeSH Terms: conditions — Breast Neoplasms | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual manoeuver + stretching (Experimental): Patients will receive a manual manoeuver treatment and education to perform stretching exercises at home.
  Interventions: Other: Manual manoeuver + stretching
- stretching exercise (Active Comparator): Patients will receive education to perform stretching exercises at home.
  Interventions: Other: stretching exercise

INTERVENTIONS:
Other: Manual manoeuver + stretching — Patients in experimental group will receive, after AWS diagnose, a manual manoeuver to snap the cord, follow by a demonstration and education of the exercise to be made at home.
  Arms: Manual manoeuver + stretching
Other: stretching exercise — Patients in control group will receive, after AWS diagnose, just a demonstration and education of the exercise to be made at home.
  Arms: stretching exercise

SUMMARY:
The aim of this study is verify the effectiveness of manual maneuver associated with stretching exercises in the treatment of Axillary Web Syndrome.

DETAILED DESCRIPTION:
Axillary Web Syndrome (AWS) is one of the short / medium-term sequela of surgical treatment for breast cancer with axillary dissection (AD) or sentinel lymph node biopsy (SLNB), with incidence reported in literature between 28% and 72%. AWS could be described as a thrombophlebitis of veno-lymph vessels due to a trauma of the region subjected to surgery, with the same characteristics of "Mondor's disease" diagnosed in post-traumatic and surgical areas where is a large presence of veno-lymphatic capillaries.

The syndrome onset occur in approximately 2-4 weeks after the surgery and its complete regression happen in 3-6 months after the onset. The clinical signs frequently described are pain and tension during movement in the axillary region, elbow, forearm and wrist, following the arm lymphatic pathway. Moreover, patients report difficulties in moving the arm into activities that require a moderate range of motion and could feel and see in the affected arm cords similar to a tendon. Even if the impairment can cause disability for a limited period of time, rehabilitation is usually advice to prevent further complications such as frozen shoulder, articular impeachment syndrome and long-term chronic pain, complications that could worsen patient's quality of life with a significant increase in costs and time to recovery.

Nowadays there are no studies in the literature that demonstrate the effectiveness of physiotherapy in AWS, with just case reports describing different treatments techniques, without a scientifically defined experimented rehabilitation protocol.

This experimental, monocentric, randomized clinical trial wants verify the effectiveness of a manual maneuver associated with stretching exercises in the treatment of AWS.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with age between 18 and 70 years old
* Axillary dissection with or without plastic reconstruction with prothesis
* Positive diagnose of axillary web syndrome.
* Patients without mental or psychological problems which could affect the proposed treatment execution.
* Signed informed consensus form.

Exclusion Criteria:

* Chronic or acute upper limb pathology which could affect the proposed treatment execution.
* Patients with mental or psychological problems which could affect the proposed treatment execution.
* Plastic reconstruction with abdominal (DIEP or TRAM) and dorsal grafts or with expander.
* Previous head and neck, sentinel lymph node biopsy or axillary dissection surgery.
* Previous breast, axillary or head and neck radiotherapy.
* Halsted mastectomy.
* Previous lymphedema.
* Bilateral axillary dissection surgery
* Physiotherapy treatment execute outside hospital during the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-07-16 (Actual); Primary Completion 2016-01-12 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Range of motion change overtime | Baseline, 7 days and 30 days after baseline measure
  Range of motion measured with a handheld goniometer, in degrees.

SECONDARY OUTCOMES:
Lymphedema assessment | 3 years after baseline measure
  Lymphedema measured with centimetric and constant dielectric method

OTHER OUTCOMES:
Pain change overtime | Baseline, 7 days and 30 days after baseline measure
  Pain measured with 0-10 numeric rate scale

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Sandrin, Principal Investigator — European Institute of Oncolgy
Locations (1):
- Istituto Europeo di Oncologia, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergmann A, Mendes VV, de Almeida Dias R, do Amaral E Silva B, da Costa Leite Ferreira MG, Fabro EA. Incidence and risk factors for axillary web syndrome after breast cancer surgery. Breast Cancer Res Treat. 2012 Feb;131(3):987-92. doi: 10.1007/s10549-011-1805-7. Epub 2011 Oct 11. PMID 21987036
- [Background] Cheville AL, Tchou J. Barriers to rehabilitation following surgery for primary breast cancer. J Surg Oncol. 2007 Apr 1;95(5):409-18. doi: 10.1002/jso.20782. PMID 17457830
- [Background] Wariss BR, Costa RM, Pereira AC, Koifman RJ, Bergmann A. Axillary web syndrome is not a risk factor for lymphoedema after 10 years of follow-up. Support Care Cancer. 2017 Feb;25(2):465-470. doi: 10.1007/s00520-016-3424-7. Epub 2016 Oct 4. PMID 27704260
- [Background] Torres Lacomba M, Mayoral Del Moral O, Coperias Zazo JL, Yuste Sanchez MJ, Ferrandez JC, Zapico Goni A. Axillary web syndrome after axillary dissection in breast cancer: a prospective study. Breast Cancer Res Treat. 2009 Oct;117(3):625-30. doi: 10.1007/s10549-009-0371-8. Epub 2009 Mar 21. PMID 19306057
- [Background] Moskovitz AH, Anderson BO, Yeung RS, Byrd DR, Lawton TJ, Moe RE. Axillary web syndrome after axillary dissection. Am J Surg. 2001 May;181(5):434-9. doi: 10.1016/s0002-9610(01)00602-x. PMID 11448437